CLINICAL TRIAL: NCT00292240
Title: Brief Youth Substance Use Intervention for Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21DA018854 (NIH)
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Consumption; Drug Abuse
Keywords: brief motivational intervention; teens; substance use
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders

INTERVENTIONS:
Behavioral: Brief motivational substance use intervention

SUMMARY:
Over the past decade, many new programs intended to prevent substance use among adolescents have been developed and evaluated. There has been a recent shift towards brief interventions for youth in school (Brown, 2001; D'Amico and Fromme, 2002) and health care settings, such as emergency rooms and inpatient clinics (Barnett et al., 2001; Colby et al., 1998; Monti et al., 1999). Although the primary care setting presents a unique opportunity to intervene with youth concerning drug use, such as marijuana or inhalants, many youth are not screened for use (Friedman et al., 1990; Johnson and Millstein, 2003; Middleman et al., 1995) and preventive services in this setting are significantly below recommended levels (Halpern-Felsher et al., 2000; Klein et al., 2001; Ozer et al., 2001). The objectives of the proposed research are to: 1) explore the feasibility of adapting a brief intervention from our previous work for use in the primary care (PC) setting, and 2) assess the short-term efficacy of the intervention in the PC setting. During year 1, focus groups of high-risk youth (n=16), parents (n=8), and providers (n=8) will provide feedback on barriers to implementing a substance use brief intervention in a PC setting. We define high-risk youth as those who may have already developed regular patterns of use or have experienced some problems due to their use. In addition, the intervention will be pilot tested with 10 high-risk youth who will provide feedback on intervention content. Revisions will be made to the intervention curriculum based on this feedback and in year 2, the short-term efficacy of the intervention will be tested with a small sample of high-risk youth (n=30). This study will extend brief intervention research for youth, as it will be one of the first to examine the feasibility of implementing a brief substance use intervention to PC with high-risk youth and to determine the impact of this intervention on short-term outcomes.

DETAILED DESCRIPTION:
Over the past decade, many new programs intended to motivate adolescents to decrease substance use have been developed and evaluated. There has been a recent shift towards brief interventions for youth in school (Brown, 2001; D'Amico and Fromme, 2002) and health care settings, such as emergency rooms and inpatient clinics (Barnett et al., 2001; Colby et al., 1998; Monti et al., 1999). Many youth who use drugs and alcohol are at risk for consequences (Johnston et al., 2003). The primary care setting presents a unique opportunity to intervene with substance abusing adolescents as 70% of youth age 10-18 visit a physician approximately 3 times a year (Gans and Newacheck, 1991; Monheit and Cunningham, 1992). However, many youth are not screened for use in this setting (Friedman et al., 1990; Johnson and Millstein, 2003; Middleman et al., 1995) and preventive services are significantly below recommended levels (Halpern-Felsher et al., 2000; Klein et al., 2001; Ozer et al., 2001). This may be due to clinician time constraints and insufficient training on substance abuse, adolescent fear that parents may see the record, and clinician discomfort in asking questions about substance use (Blum, 1987; Blum et al., 1996; Lustig et al., 2001; Marcell et al., 2002; Middleman et al., 1995).

The present proposal is designed to meet the objectives of the Exploratory/Developmental Grants program (R21) for studies that will contribute to the development of future, more intensive and larger research programs. The objectives of the proposed research are to: 1) explore the feasibility of adapting a brief intervention from our previous work in schools and emergency rooms for use in the primary care setting, and 2) assess the short-term efficacy of the intervention in the primary care setting. This project serves as our first step in an innovative line of research designed to examine the viability of utilizing brief interventions targeting adolescent drug use in primary care settings. Our objectives will be accomplished through the following aims:

1. Explore the feasibility of adapting a brief intervention for high-risk youth in a primary care (PC) setting. We will determine barriers and facilitative factors associated with implementing a brief intervention in a PC setting through focus groups with high-risk youth (n=16), parents (n=8), and clinicians (n=8). Intervention content will be established through modifications of our previous brief intervention work in school and hospital settings and from focus group feedback from adolescents, clinicians, and parents. We anticipate the intervention will take 15 minutes and will be implemented by a clinician (e.g., nurse) in the PC setting. The intervention will emphasize motivational techniques and will address a variety of substances, including marijuana, inhalants, alcohol, and cigarettes. We will pilot test the intervention with a small sample of high-risk youth (n=10) to obtain feedback to discern whether the intervention was difficult to implement (e.g., time constraints, comfort level) and how youth felt about receiving feedback from their clinicians on their substance use (e.g., was it helpful? What other topics would they have liked to discuss?). We will modify content based on this feedback.
2. Implement and assess short-term efficacy of a brief intervention for high-risk youth in a PC setting. We will implement the intervention in the PC setting with a small sample of high-risk youth (n=30) and assess its potential impact on short-term outcomes (e.g., perceived prevalence of peer use, self-change efforts) at a 3-month follow up. These youth will be compared to an assessment only control group (n=30).

This research will culminate with the development of a longer-term plan for implementing and evaluating the intervention more intensively with a larger sample. Products will include: 1) intervention materials adapted for use with high-risk youth in primary care settings, 2) pilot data on intervention feasibility and implementation, and 3) an R01 application to examine the generalizability and long-term impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years old
* english speaker
* screen positive for alcohol and/or drug use

We use a brief screener to identify youth at high-risk for drug or alcohol abuse. The CRAFFT was developed by Knight and colleagues to screen youth for alcohol and other drug use and is a mnemonic based on the six questions it asks. The CRAFFT is comprised from items from the RAFFT (Riggs and Alario, 1989), DAP (Drug and Alcohol Problems) (Klitzner et al., 1987) and POSIT (Problem Oriented Screening Instrument for Teenagers) (Rahdert, 1991). The CRAFFT is brief, highly correlated with the Personal Involvement with Chemicals Scale (PICS), a criterion standard (r = .84), and is practical for use in a primary care setting as it takes only a few minutes to administer (Knight et al., 1999). The measure includes the following Yes/No questions: 1) have you ever ridden in a car driven by someone (including yourself) who was high or had been using alcohol or drugs?, 2) do you ever use alcohol or drugs to relax, feel better about yourself, or fit in?, 3) do you ever use alcohol or drugs while you are by yourself (alone)?, 4) do you ever forget things you did while using alcohol or drugs?, 5) have you ever gotten into trouble while you were using alcohol or drugs?, and 6) do your family and friends ever tell you that you should cut down on your drinking or drug use?. The six items have a cut-off score of 2 or greater with a sensitivity of 92.3% and specificity of 82.5% for long-term treatment need (as identified by PICS scores) (Knight et al., 1999). We use a cut-off of 1 or greater, reflecting a less stringent criterion for "high-risk" that includes adolescents with potential problems who could benefit from a brief intervention in the primary care setting.

Exclusion Criteria:

* spanish speaker
* outside of age range
* does not qualify on screening questionnaire as using alcohol and/or drugs

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2004-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
alcohol, tobacco, drug use
alcohol and drug consequences
self-change efforts
perceived peer use
positive and negative outcome expectancies
all measures taken at pre intervention and 3 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. D'Amico, Ph.D., Principal Investigator — RAND
Locations (1):
- Los Angeles Free Clinic, Los Angeles, California, United States